CLINICAL TRIAL: NCT03564275
Title: Assessing the Effectiveness of Photon Therapy With a Proton Therapy Boost in the Treatment of Prostate Cancer as Compared to Photon Therapy Alone
Brief Title: Proton Boost in Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, William Barrett, Director, University of Cincinnati Cancer Institute Medical Director, Charles M. Barrett Cancer Center Professor and Chairman, Radiation Oncology University of Cincinnati, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1091
Record Dates: First submitted 2018-05-18; First posted 2018-06-20 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cancer of the Prostate
Keywords: Radiation Therapy; Proton Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Matched pair analysis. Each prospective patient will be matched with two historical patients based on the inclusion, exclusion and match criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective Treatment Group (Experimental): Proton Boost
  Interventions: Radiation: Proton Boost
- Retrospective Comparison Group (No Intervention): Retrospective patients previously treated with standard of care photon therapy. There is no patient interaction with this group. Data collection from medical records only.

INTERVENTIONS:
Radiation: Proton Boost — 13-15 treatments with proton therapy given as a boost to standard of care photon therapy
  Arms: Prospective Treatment Group

SUMMARY:
This study uses photon radiation with a proton boost to treat prostate cancer. The purpose of this study is to determine if proton therapy as a boost following photon intensity modulated radiation therapy (IMRT) produces decreased toxicity as compared to conventional photon IMRT alone in the treatment of prostate cancer. Our secondary objective is to determine the effectiveness of this treatment regimen. Effectiveness will be determined by length of time to progression or recurrence of disease and overall survival. Patients on this study will be treated with a course of photon radiation therapy followed by a boost course of proton radiation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosis of low risk prostate cancer (T1c-T2a, Gleason 6, Prostate Specific Antigen (PSA) <10) -OR-
* Diagnosis of intermediate risk prostate cancer (T1c-T2c, Gleason 7 and/or PSA 10- 20)
* Life expectancy >10 yrs
* Physically and mentally capable of signing the consent form of their own volition

Exclusion Criteria:

* < 18 years of age
* Diagnosis of high risk prostate cancer (T3 or higher, Gleason >7 and/or PSA >20)
* Current or historical use of androgen deprivation therapy
* Nodal positivity
* Previous cancer excluding non-melanoma skin cancer
* History of prostatectomy
* History of brachytherapy for prostate cancer
* Life expectancy <10 yrs
* Physically or mentally incapable of signing the consent form of their own volition

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2033-04 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Hematuria - Change from baseline | Post therapy - 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months, 6,7,8,9,10 years
  Common Terminology Criteria for Adverse Events - Hematuria Scale - 1(least severe) - 5 (most severe)
Urinary Incontinence - Change from baseline | Post therapy - 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months, 6,7,8,9,10 years
  Common Terminology Criteria for Adverse Events - Urinary Incontinence Scale - 1(least severe) - 3 (most severe)
Dysuria - Change from baseline | Post therapy - 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months, 6,7,8,9,10 years
  Presence or Absence
International Prostate Symptom Score - Change from baseline | Post therapy - 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months, 6,7,8,9,10 years
  Records patient reported urinary symptoms - Scale 1-35 - 1-7 Mild symptoms, 8-19 Moderate symptoms, 20-35 Severe symptoms
Rectal Bleeding - Change from baseline | Post therapy - 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months, 6,7,8,9,10 years
  Common Terminology Criteria for Adverse Events - Rectal Hemorrhage Scale - 1(least severe) - 5 (most severe)
Erectile Dysfunction - Change from baseline | Post therapy - 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54, 60 months, 6,7,8,9,10 years
  Common Terminology Criteria for Adverse Events - Erectile Dysfunction Scale - 1(least severe) - 3 (most severe)

SECONDARY OUTCOMES:
Progression Free Survival | Monitored for 10 years after completion of radiation therapy
  Measured by time to cancer recurrence
Overall Survival | Monitored for 10 years after completion of radiation therapy
  Measured by time to cancer-related death

CONTACTS AND LOCATIONS:
Overall Officials: William Barrett, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Boccon-Gibod LM, Dumonceau O, Toublanc M, Ravery V, Boccon-Gibod LA. Micro-focal prostate cancer: a comparison of biopsy and radical prostatectomy specimen features. Eur Urol. 2005 Dec;48(6):895-9. doi: 10.1016/j.eururo.2005.04.033. PMID 16125298
- [Background] Gregori A, Vieweg J, Dahm P, Paulson DF. Comparison of ultrasound-guided biopsies and prostatectomy specimens: predictive accuracy of Gleason score and tumor site. Urol Int. 2001;66(2):66-71. doi: 10.1159/000056573. PMID 11223746
- [Background] Scales CD, Amling CL, Kane CJ, et al. Can unilateral Prostate Cancer be Reliably Predicted Based Upon Biopsy Features? J Urol. 2006; 175:373.
- [Background] Schulte RT, Wood DP, Daignault S, Shah RB, Wei JT. Utility of extended pattern prostate biopsies for tumor localization: pathologic correlations after radical prostatectomy. Cancer. 2008 Oct 1;113(7):1559-65. doi: 10.1002/cncr.23781. PMID 18726951
- [Background] Arrayeh E, Westphalen AC, Kurhanewicz J, Roach M 3rd, Jung AJ, Carroll PR, Coakley FV. Does local recurrence of prostate cancer after radiation therapy occur at the site of primary tumor? Results of a longitudinal MRI and MRSI study. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):e787-93. doi: 10.1016/j.ijrobp.2011.11.030. Epub 2012 Feb 11. PMID 22331003
- [Background] Pollack A, Zagars GK, Starkschall G, Antolak JA, Lee JJ, Huang E, von Eschenbach AC, Kuban DA, Rosen I. Prostate cancer radiation dose response: results of the M. D. Anderson phase III randomized trial. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1097-105. doi: 10.1016/s0360-3016(02)02829-8. PMID 12128107
- [Background] Peeters ST, Heemsbergen WD, Koper PC, van Putten WL, Slot A, Dielwart MF, Bonfrer JM, Incrocci L, Lebesque JV. Dose-response in radiotherapy for localized prostate cancer: results of the Dutch multicenter randomized phase III trial comparing 68 Gy of radiotherapy with 78 Gy. J Clin Oncol. 2006 May 1;24(13):1990-6. doi: 10.1200/JCO.2005.05.2530. PMID 16648499
- [Background] Andrzejewski P, Kuess P, Knausl B, Pinker K, Georg P, Knoth J, Berger D, Kirisits C, Goldner G, Helbich T, Potter R, Georg D. Feasibility of dominant intraprostatic lesion boosting using advanced photon-, proton- or brachytherapy. Radiother Oncol. 2015 Dec;117(3):509-14. doi: 10.1016/j.radonc.2015.07.028. Epub 2015 Sep 6. PMID 26349588
- [Background] Bossart EL, Stoyanova R, Sandler K, Studenski M, Orman A, Abramowitz M, Pollack A. Feasibility and Initial Dosimetric Findings for a Randomized Trial Using Dose-Painted Multiparametric Magnetic Resonance Imaging-Defined Targets in Prostate Cancer. Int J Radiat Oncol Biol Phys. 2016 Jun 1;95(2):827-34. doi: 10.1016/j.ijrobp.2016.01.052. Epub 2016 Feb 4. PMID 27020109
- [Background] Johansson S, Astrom L, Sandin F, Isacsson U, Montelius A, Turesson I. Hypofractionated proton boost combined with external beam radiotherapy for treatment of localized prostate cancer. Prostate Cancer. 2012;2012:654861. doi: 10.1155/2012/654861. Epub 2012 Jul 8. PMID 22848840
- [Background] Nihei K, Ogino T, Ishikura S, Kawashima M, Nishimura H, Arahira S, Onozawa M. Phase II feasibility study of high-dose radiotherapy for prostate cancer using proton boost therapy: first clinical trial of proton beam therapy for prostate cancer in Japan. Jpn J Clin Oncol. 2005 Dec;35(12):745-52. doi: 10.1093/jjco/hyi193. Epub 2005 Nov 28. PMID 16314345